CLINICAL TRIAL: NCT05805371
Title: A Phase 1b Study Evaluating Combinations With PSCA-Targeting Chimeric Antigen Receptor (CAR)-T Cells for Patients With PSCA+ Metastatic Castration-Resistant Prostate Cancer
Brief Title: PSCA-Targeting CAR-T Cells Plus or Minus Radiation for the Treatment of Patients With PSCA+ Metastatic Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22378; NCI-2023-02186 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22378 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-03-24; First posted 2023-04-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy; Specimen Handling; Radiation; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment plan I (PSCA CAR T-cells) (Experimental): Patients undergo leukapheresis and lymphodepletion and receive PSCA-CAR T cells IV up to 3 times on study. Patients undergo bone scan, CT scan, tumor biopsy, and collection of blood, stool, and urine samples throughout the trial.
  Interventions: Biological: Autologous Anti-PSCA-CAR-4-1BB/TCRzeta-CD19t-expressing T-lymphocytes; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Leukapheresis; Procedure: Lymphodepletion Therapy
- Treatment plan II (PSCA CAR T-cells, radiation) (Experimental): Patients undergo leukapheresis, radiation in 2 doses, and lymphodepletion, and receive PSCA-CAR T cells IV up to 3 times on study. Patients undergo bone scan, CT scan, tumor biopsy, and collection of blood, stool, and urine samples throughout the trial.
  Interventions: Biological: Autologous Anti-PSCA-CAR-4-1BB/TCRzeta-CD19t-expressing T-lymphocytes; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Radiation: External Beam Radiation Therapy; Procedure: Leukapheresis; Procedure: Lymphodepletion Therapy

INTERVENTIONS:
Biological: Autologous Anti-PSCA-CAR-4-1BB/TCRzeta-CD19t-expressing T-lymphocytes — Given IV
  Other Names: Autologous Anti-PSCA(dCH2)BBz-CAR T-cells; Autologous Anti-PSCA-CAR-4-1BB/TCRzeta-CD19t-expressing T-cells; PSCA(dCH2)BBzeta-CAR T-cells
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood, stool, and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Radiation: External Beam Radiation Therapy — Undergo radiation
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
  Arms: Treatment plan II (PSCA CAR T-cells, radiation)
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Procedure: Lymphodepletion Therapy — Undergo lymphodepletion
  Other Names: Lymphodepleting Therapy; Lymphodepletion

SUMMARY:
This phase Ib trial tests the safety, side effects, and best dose of autologous anti-prostate stem cell antigen (PSCA)-chimeric antigen receptor (CAR)-4-1BB/TCRzeta-CD19t-expressing T-lymphocytes (PSCA-CAR T cells), plus or minus radiation, in treating patients with castration-resistant prostate cancer that has spread from where it first started (primary site) to other places in the body (metastatic). Castration-resistant prostate cancer continues to grow and spread despite the surgical removal of the testes or medical intervention to block androgen production. CAR T-cell therapy is a type of treatment in which a patient's T cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. T cells are taken from a patient's blood. Then the gene for a special receptor that binds to a certain protein on the patient's cancer cells is added to the T cells in the laboratory. The special receptor is called a chimeric antigen receptor (CAR). Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers. Radiation therapy uses high energy x-rays to kill cancer cells and shrink tumors. Giving PSCA-targeting CAR T-cells, with or without radiation, may kill more tumor cells in men with castration-resistant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the feasibility, safety, and activity of lymphodepleting chemotherapy followed by up to 3 cycles of 50M PSCA-CAR T cell immunotherapy per course either alone (treatment plan 1 [TP1]) or in combination with metastasis-directed radiation therapy (MDRT) (treatment plan 2 [TP2]) in adult patients with metastatic castration-resistant prostate cancer (mCRPC).

SECONDARY OBJECTIVES:

I. Describe persistence and expansion of CAR T cells in peripheral blood (PB). II. Describe cytokine levels over the study period. III. Estimate disease response rates. IV. Estimate 6-month progression-free survival (PFS) rate. V. Estimate 1-year overall survival (OS) rate.

EXPLORATORY OBJECTIVES:

I. Describe the immune landscape changes in PB and tumors. II. Describe phenotype of CAR T cells in PB. III. Describe tumor evolution in PB (circulating tumor cells [CTCs], circulating cell-free deoxyribonucleic acid [DNA] [cfDNA]) and tumors.

IV. Determine whether urine cytokines and cellularity is predictive of cystitis occurrence/severity.

V. Analyze microbial changes in stool associated with CAR T cell therapy.

OUTLINE: Patients are assigned to 1 of 2 treatment plans.

TREATMENT PLAN I: Patients undergo leukapheresis and lymphodepletion and receive PSCA-CAR T cells intravenously (IV) up to 3 times on study.

TREATMENT PLAN II: Patients undergo leukapheresis, radiation in 2 doses, and lymphodepletion, and receive PSCA-CAR T cells IV up to 3 times on study.

Patients in both arms undergo bone scan, computed tomography (CT) scan, tumor biopsy, and collection of blood, stool and urine samples throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative (brown)

  * Assent, when appropriate, will be obtained per institutional guidelines

    * Note: For research participants who do not speak English, a short form consent may be used with a City of Hope (COH) certified interpreter/translator to proceed with screening and leukapheresis, while the request for a translated main consent is processed. However, the research participant is allowed to proceed with lymphodepletion and CAR T cell infusion only after the translated main consent form is signed
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 or Karnofsky Performance Status (KPS) >= 70%
* Documented castration resistant prostate cancer (mCRPC) (Note: castration will be defined by a testosterone < 50 ng/dL achieved by orchiectomy or luteinizing hormone-releasing hormone [LHRH] agonist/antagonist therapy)

  * Documented PSCA+ tumor expression as evaluated by the COH Pathology Clinical Trials Specimen Qualification Laboratory (CTSQL)

    * Fresh or archival biopsy samples may be tested for PSCA expression during screening for eligibility purposes. The results from soft tissue biopsies will be used to confirm eligibility for participants who have a soft-tissue lesion biopsy obtained, but bone biopsy staining results will not impact eligibility since immunohistochemistry (IHC) staining for PSCA has not been optimized in bone specimens. Subjects who undergo bone biopsy on study will be qualified based on the archival tissue result
  * Progression of disease manifest by one of the following means during treatment with at least one advanced androgen targeted therapy (e.g., abiraterone or enzalutamide):

    * Rising prostate specific antigen (PSA) documented on 2 occasions at least 7 days apart, with absolute increase > 2 ng/dL despite testosterone < 50 OR
    * Radiographic evidence of new metastatic foci on CT or bone scan, or soft tissue progression by Response Evaluation Criteria in Solid Tumors (RECIST)
  * For treatment plan 2, subjects must have at least one and up to 3 metastatic lesions which have not previously been radiated and which is safe for treatment with radiation 16 gray (Gy) in 2 fractions
* Fully recovered from the acute toxic effects (except alopecia) to =< grade 1 to prior anti-cancer therapy
* If there has been prior chemotherapy, at least 2 weeks must have elapsed prior to leukapheresis
* Prior radiotherapy is allowed provided it was not administered to the only evaluable site of disease and was completed > 14 days prior to leukapheresis
* No known contraindications to leukapheresis, steroids or tocilizumab
* Absolute neutrophil count (ANC) >= 1,000/mm^3 (within 42 days prior to enrollment)

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment
* Platelets >= 100,000/mm^3 (within 42 days prior to enrollment) NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment
* Total serum bilirubin =< 2.0 mg/dL (within 42 days prior to enrollment)

  * Patients with Gilbert syndrome may be included if their total bilirubin is =< 3.0 x upper limit of normal (ULN) and direct bilirubin =< 1.5 x ULN
* Aspartate aminotransferase (AST) =< 2.5 x ULN (within 42 days prior to enrollment)
* Alanine aminotransferase (ALT) =< 2.5 x ULN (within 42 days prior to enrollment)
* Creatinine clearance of >= 50 mL/min per 24 hour urine test or the Cockcroft-Gault formula (within 42 days prior to enrollment)
* Corrected QT interval (QTc) =< 480 ms

  * Note: to be performed within 28 days prior to day 1 of protocol therapy
* Cardiac function (12 lead- electrocardiogram [ECG]) without acute abnormalities requiring investigation or intervention (within 42 days prior to enrollment)
* Seronegative for human immunodeficiency virus (HIV) antigen (Ag)/antibody (Ab) combo, hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative), and syphilis (rapid plasma reagin [RPR])

  * If positive, hepatitis C ribonucleic acid (RNA) quantitation must be performed OR
  * If seropositive for HIV, HCV or HBV, nucleic acid quantitation must be performed. Viral load must be undetectable
  * Note infectious disease testing to be performed within 28 days prior to day 1 of protocol therapy
* Meets other institutional and federal requirements for infectious disease titer requirements

  * Note Infectious disease testing to be performed within 28 days prior to day 1 of protocol therapy
* Agreement by males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 3 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized

Exclusion Criteria:

* Concurrent use of systemic steroids or chronic use of immunosuppressant medications. Recent or current use of inhaled steroids is not exclusionary. Physiologic replacement of steroids (prednisone =< 7.5 mg /day, or hydrocortisone =< 20 mg /day) is allowed
* Subjects with clinically significant arrhythmia or arrhythmias not stable on medical management within two weeks of screening
* Subjects with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system, including seizure disorder
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia
* History of stroke or intracranial hemorrhage within 6 months prior to screening
* History of other malignancies, except for malignancy surgically resected (or treated with other modalities) with curative intent, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin; non-muscle invasive bladder cancer; malignancy treated with curative intent with no known active disease present for >= 3 years
* Clinically significant uncontrolled illness
* Active infection requiring antibiotics
* Known history of immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2028-11-11 (Estimated); Study Completion 2028-11-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Post chimeric antigen receptor (CAR) T cell infusion up to 15 years
  Dose limiting toxicities (DLTs), cystitis, grade 3 toxicities and the full toxicity profile as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events version 5 and cytokine release syndrome (CRS) and neurotoxicity as assessed by modified CRS grading. The recommended phase 2 dose (RP2D) will be based on the treatment plan 2 toxicity, activity and correlative data. Rates and associated 90% Clopper and Pearson binomial confidence limits will be estimated for DLTs within the DLT period. Tables will be created to summarize all toxicities and side effects by attribution to treatment arm, dose, organ and severity.
50% prostate specific antigen (PSA) level reduction | From baseline measurement up to 1 year post study treatment
  Statistical and graphical methods will be used to describe cytokine levels (peripheral blood) and PSA levels over the study period.

SECONDARY OUTCOMES:
Persistence of CAR T cells | Up to 28 days post last study treatment
  Maximum persistence (in days) will be described by treatment plan, recognizing the number of CAR T cycles the participant received.
Expansion of CAR T cells | Up to 28 days post last study treatment
  Peak expansion (log10 copies/ug of genomic deoxyribonucleic acid [DNA]) will be described by treatment plan, recognizing the number of CAR T cycles the participant received.
PSCA tumor expression | From baseline to end of cycle 1 (Cycle length is 56 days)
  PSCA expression on tumor cells by IHC and/or flow cytometry.
Serum cytokine profile | Before CAR T cell infusion through completion of cycle 2, up to 4 months (Cycle length is 56 days)
  Statistical and graphical methods will be used.
Overall survival | From time of lymphodepletion to date of death, assessed at 1 year
  Rates and associated 90% Clopper and Pearson binomial confidence limits will be estimated.
Progression-free survival | Survival without radiographic evidence of disease progression from time of lymphodepletion to the date of progression or death, assessed at 6 months
  Rates and associated 90% Clopper and Pearson binomial confidence limits will be estimated.
Disease response by PSA | From baseline up to 1 year post study treatment
  Rates and associated 90% Clopper and Pearson binomial confidence limits will be estimated.
Disease response by immune-modified Response Evaluation Criteria in Solid Tumors criteria | At baseline, and months 3, 6, 9 and 12
  Rates and associated 90% Clopper and Pearson binomial confidence limits will be estimated.
Disease response by Prostate Cancer Working Group criteria | At baseline, and months 3, 6, 9 and 12
  Rates and associated 90% Clopper and Pearson binomial confidence limits will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya B Dorff, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States